CLINICAL TRIAL: NCT01736930
Title: Reduction of Nocturnal Hypoglycemia by Using Predictive Algorithms and Pump Suspension: An Outpatient Pilot Feasibility and Safety Study
Brief Title: An Outpatient Pump Shutoff Pilot Feasibility and Safety Study
Acronym: PSO1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PSO1; R01DK085591 (NIH)
Record Dates: First submitted 2012-11-20; First posted 2012-11-29 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Hypoglycemia; Continuous Glucose Monitoring; Pump Suspension
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Predictive pump suspension algorithm (Active Comparator): The study laptop will be running actively during the night and suspending the patient's pump if the algorithm predicts hypoglycemia based on the patient's continuous glucose sensor trend.
  Interventions: Device: Pump suspension
- Standard of Care (No Intervention): The control algorithm will run passively and not recommend suspensions or resumption to the patient's pump.

INTERVENTIONS:
Device: Pump suspension — The study laptop will communicate to the pump causing suspension based on output from the algorithm which predicts hypoglycemia based on the continuous glucose sensor trend.
  Arms: Predictive pump suspension algorithm

SUMMARY:
The purpose of this study is to evaluate an overnight system that will turn off the insulin pump automatically if the system predicts that a low blood sugar is likely. The study system includes a combination continuous glucose monitor (CGM)/ insulin pump made by Medtronic MiniMed, Inc and a regular laptop computer that runs a computer program that predicts low blood sugar. It works by (1) measuring the glucose levels under the skin with a continuous glucose monitor, (2) using a computer program on a laptop to predict what will happen to the glucose level over the next 35-55 minutes, and (3) turning off the insulin pump when the computer program predicts that low blood sugar will occur. We have tested this system overnight in the hospital and are ready to test the system in the home environment to learn more about how well it will work and to make sure that the blood sugar does not go too high when the pump shuts off.

This study has several phases and will take about a month or a little more for a patient to complete. Patients will use the study system for about 5 days at home to show that the patient is able to use it correctly. After that, the patient will be asked to use the study system each night for an additional 3-4 weeks. During this time, the system will be active for two-thirds of the nights and not active for one-third of the nights. When the system is active and predicts that your blood sugar will become low, the insulin pump will shut off for up to 2 hours.

The study will include 2 clinical centers in the United States.

DETAILED DESCRIPTION:
Patients who meet all eligibility criteria will use the study system overnight at home for about 5 nights to demonstrate their ability to use the system and submit study data to the Coordinating Center.

Patients who successfully demonstrate their ability to use the system as described above will be eligible for the randomized trial phase. This phase consists of use of the full system as an outpatient for approximately 21 nights:

* Each night the blood glucose level will be checked with the study blood glucose (BG) meter and used to perform a calibration of the CGM. The calibration must occur no more than 90 minutes prior to activation of the system. NOTE: Patients will be instructed to calibrate the CGM per manufacturer guidelines.
* Then the system will be activated, linking the CGM and insulin pump to the computer at the bedside.
* A randomization schedule on the laptop will be used to determine whether the 'pump shut off' application will be active that night or not.
* Patients will be blinded as to whether the pump shut off is active when a session is initiated each night.
* There will not be an alarm if the pump shuts off. The CGM alarm will be set to 60 mg/dL. When a CGM alarm occurs, the patient will be asked to measure the blood glucose with a BG meter, if he/she is aware of the alarm.
* The time period for outcome assessment each night will be from the time the system is activated until it is turned off in the morning.
* Pump shut off, when it occurs, will be for up to 2 hours. Multiple instances of pump suspension can occur if there are recurrent predictions of hypoglycemia during the night.
* Patients will be asked to check blood glucose with the study BG meter, blood ketones with the study ketone meter, and urine ketones with a ketone strip each morning prior to breakfast and enter the results on the study laptop. The patient will be instructed to contact the study physician if the blood glucose or ketone readings are out of an expected range. Patients will be contacted if these morning safety values are not reported as required or are out of range.
* Patients will be asked to record all overnight carbohydrate intake on the study laptop.
* Patients will be asked to perform periodic data uploads using the study laptop. Monitoring processes will ensure that the patient is contacted if these uploads do not occur as required, or if review of an upload reveals any extreme, prolonged episodes of low or high blood glucose readings, or elevated morning blood glucose, blood ketone, or urine ketone values.

Upon completion of the study, patients as well as study clinicians will be asked to complete a questionnaire regarding use of the study system.

There will a follow-up visit after completion of 21 successful nights of study system use. A successful night of study system use is defined as use of the system for at least four hours. Phone contacts with the patients will be made once a week.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year and an insulin infusion pump for at least 6 months
* Age >=18.0 years
* HbA1c <=8.0%
* Availability of internet access for periodic upload of study data
* Experience using the Medtronic pump and CGM and investigator is confident that subject will use CGM on a near-daily basis during the study
* Nocturnal hypoglycemia meeting the following criterion based on CGM download: during the most recent 15 nights with CGM glucose data (must be within the past 42 days), one or more nights with a sensor glucose value <=70 mg/dL.

Exclusion Criteria:

* Diabetic ketoacidosis in the past 3 months
* Hypoglycemic seizure or loss of consciousness in the past 6 months
* History of seizure disorder (except for hypoglycemic seizure)
* Coronary artery disease or heart failure
* Cystic fibrosis
* Current use of oral/inhaled glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
* History of ongoing renal disease (other than microalbuminuria). Creatinine level to have been obtained within the last year if subject has diabetes of >10 years duration or is over 50 years of age. If creatinine is > 1.5 mg/dL, the subject is excluded.
* History of liver disease
* Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as: inpatient psychiatric treatment in the past 6 months, uncontrolled adrenal disorder, and/or abuse of alcohol
* Pregnancy: A negative urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Buckingham, MD, Study Chair — Stanford University; Roy W Beck, MD, PhD, Principal Investigator — Jaeb Center for Health Research; John Lum, MS, Study Director — Jaeb Center for Health Research
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado

REFERENCES:
- [Result] Buckingham BA, Cameron F, Calhoun P, Maahs DM, Wilson DM, Chase HP, Bequette BW, Lum J, Sibayan J, Beck RW, Kollman C. Outpatient safety assessment of an in-home predictive low-glucose suspend system with type 1 diabetes subjects at elevated risk of nocturnal hypoglycemia. Diabetes Technol Ther. 2013 Aug;15(8):622-7. doi: 10.1089/dia.2013.0040. Epub 2013 Jul 24. PMID 23883408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at Stanford University and the Barbara Davis Center. A total of 20 subjects were enrolled between January 1, 2012 and June 30, 2012. Nineteen participants 18-56 years old with type 1 diabetes (HbA1c 6.0%-7.7%) completed the trial.
Pre-assignment Details: After the run-in phase, a 21-night randomized trial was conducted in which each night was randomly assigned 2:1 to have either the predictive low glucose suspend system active (intervention) or inactive (control). Participants were current users of the MiniMed Paradigm® REAL-Time Revel™ System and Sof-sensor® glucose sensor at time of enrollment.
Groups:
- Randomized Nights- Treatment or Control: Each study night will be randomized to have either Predictive Low Glucose Suspend or to be inactive (control). On nights randomized to the intervention treatment, the study laptop will be running actively during the night and suspending the patient's pump if the algorithm predicts hypoglycemia based on the patient's continuous glucose sensor trend. (Pump suspension : The study laptop will communicate to the pump causing suspension based on output from the algorithm which predicts hypoglycemia based on the continuous glucose sensor trend.) On control nights, the algorithm will run passively and not recommend suspensions or resumption to the patient's pump.
Period: Overall Study
Arm/Group | Randomized Nights- Treatment or Control
Started | 20 (Each night randomized to have either Predictive Low Glucose suspend or inactive (control).)
Completed | 19 (Each night randomized to have either Predictive Low Glucose suspend or inactive (control).)
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Each night randomized to have either Predictive Low Glucose suspend or inactive (control).
Arm/Group | Randomized Nights- Treatment or Control
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Morning Blood Glucose (mg/dL)- Algorithm 1
Description: The primary safety outcome will be evaluated by comparing the intervention and control nights and nights with vs. without actual shut-off of the pump for several measures of hyperglycemia such as mean morning blood glucose (mg/dL).
  An objective was to evaluate and refine the control algorithm. The data were reviewed periodically during the study with the pre-stated goal of determining whether any changes should be made in the control algorithm. Algorithm 1 was used for the first 105 nights of the study (38 Control nights and 67 Intervention nights). The horizon prediction time of algorithm 1 was set at 70 minutes.
Time Frame: 21 study nights
Measure: Mean (Standard Deviation); unit: mg/dl
Units Other Than Participants: Number of Mornings Analyzed
Groups:
- Predictive Pump Suspension Algorithm: The study laptop will be running actively during the night and suspending the patient's pump if the algorithm predicts hypoglycemia based on the patient's continuous glucose sensor trend.
  Pump suspension : The study laptop will communicate to the pump causing suspension based on output from the algorithm which predicts hypoglycemia based on the continuous glucose sensor trend.
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 5 | 5
Number analyzed (Number of Mornings Analyzed) | 67 | 38
mg/dl | 158 (52) | 125 (53)

2. Primary Outcome: Mean Morning Blood Glucose (mg/dL)- Algorithm 2
Description: The primary safety outcome will be evaluated by comparing the intervention and control nights and nights with vs. without actual shut-off of the pump for several measures of hyperglycemia such as mean morning blood glucose (mg/dL).
  Algorithm 1 was modified to reduce the hypoglycemia prediction horizon from 70 minutes to 50 minutes, to suspend the pump only when the continuous glucose monitor sensor glucose value was ≤ 230 mg/dl, not suspend if there was a drop of >40 mg/dl in consecutive sensor glucose readings, and to resume insulin delivery at the first rise in sensor glucose following a suspension. There was 156 nights of study data collected (48 Control nights and 108 Intervention nights) using algorithm 2.
Time Frame: 21 study nights
Measure: Mean (Standard Deviation); unit: mg/dl
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 12 | 10
Number analyzed (Number of Mornings Analyzed) | 108 | 48
mg/dl | 151 (57) | 138 (63)

3. Primary Outcome: Mean Morning Blood Glucose (mg/dL)- Algorithm 3
Description: The primary safety outcome will be evaluated by comparing the intervention and control nights and nights with vs. without actual shut-off of the pump for several measures of hyperglycemia such as mean morning blood glucose (mg/dL).
  The hypoglycemia prediction horizon was reduced further in algorithm 3 to 30 minutes. A total of 114 study nights (37 Control nights and 77 Intervention nights) using algorithm 3.
Time Frame: 21 study nights
Measure: Mean (Standard Deviation); unit: mg/dl
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 9 | 8
Number analyzed (Number of Mornings Analyzed) | 77 | 37
mg/dl | 144 (48) | 133 (57)

4. Primary Outcome: Percent Morning Blood Glucose >250 mg/dL - Algorithm 1
Description: The primary safety outcome will be evaluated by comparing the intervention and control nights and nights with vs. without actual shut-off of the pump for several measures of hyperglycemia such as the overall percentage of mornings glucose measured with home glucose meter >250 mg/dL.
Time Frame: 21 days
Measure: Number; unit: percentage of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 5 | 5
Number analyzed (Number of Mornings Analyzed) | 67 | 38
percentage of mornings | 3 | 3

5. Secondary Outcome: Mean Sensor Glucose Overnight - Algorithm 1
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 21 nights of system use
Measure: Mean (Standard Deviation); unit: mg/dl
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 5 | 5
Number analyzed (Number of Nights Analyzed) | 67 | 38
mg/dl | 158 (34) | 145 (42)

6. Secondary Outcome: Mean Sensor Glucose Overnight - Algorithm 2
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 21 nights of system use
Measure: Mean (Standard Deviation); unit: mg/dl
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 12 | 10
Number analyzed (Number of Nights Analyzed) | 108 | 48
mg/dl | 137 (36) | 123 (40)

7. Secondary Outcome: Mean Sensor Glucose Overnight - Algorithm 3
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 21 nights of system use
Measure: Mean (Standard Deviation); unit: mg/dl
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 9 | 8
Number analyzed (Number of Nights Analyzed) | 77 | 37
mg/dl | 148 (42) | 133 (37)

8. Secondary Outcome: Percentage of Sensor Glucose Values 71 to 180 mg/dL - Algorithm 1
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 21 nights of system use
Measure: Median (Inter-Quartile Range); unit: percentage of sensor glucose values
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 5 | 5
Number analyzed (Number of Nights Analyzed) | 67 | 38
percentage of sensor glucose values | 71 [51 to 91] | 76 [46 to 100]

9. Secondary Outcome: Percentage of Sensor Glucose Values 71 to 180 mg/dL - Algorithm 2
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 21 nights of system use
Measure: Median (Inter-Quartile Range); unit: percentage of sensor glucose values
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 12 | 10
Number analyzed (Number of Nights Analyzed) | 108 | 48
percentage of sensor glucose values | 90 [65 to 100] | 91 [68 to 100]

10. Secondary Outcome: Percentage of Sensor Glucose Values 71 to 180 mg/dL - Algorithm 3
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 21 nights of system use
Measure: Median (Inter-Quartile Range); unit: percentage of sensor glucose values
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 9 | 8
Number analyzed (Number of Nights Analyzed) | 77 | 37
percentage of sensor glucose values | 89 [50 to 100] | 94 [69 to 100]

11. Primary Outcome: Percent Morning Blood Glucose >250 mg/dL - Algorithm 2
Description: The primary safety outcome will be evaluated by comparing the intervention and control nights and nights with vs. without actual shut-off of the pump for several measures of hyperglycemia such as overall percentage of mornings glucose measured with home glucose meter >250 mg/dL.
Time Frame: 21 days
Measure: Number; unit: percentage of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 12 | 10
Number analyzed (Number of Mornings Analyzed) | 108 | 48
percentage of mornings | 6 | 8

12. Primary Outcome: Percent Morning Blood Glucose >250 mg/dL - Algorithm 3
Description: as for outcome 11
Time Frame: 21 days
Measure: Number; unit: percentage of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 9 | 8
Number analyzed (Number of Mornings Analyzed) | 77 | 37
percentage of mornings | 1 | 3

13. Primary Outcome: Mornings With Blood Ketones >0.6 mmol/L - Algorithm 1
Description: The primary safety outcome will be evaluated by comparing the intervention and control nights and nights with vs. without actual shut-off of the pump for several measures of hyperglycemia such as number of mornings with blood ketones >0.6 mmol/L.
Time Frame: 21 days
Measure: Number; unit: number of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 5 | 5
Number analyzed (Number of Mornings Analyzed) | 67 | 38
number of mornings | 0 | 0

14. Primary Outcome: Mornings With Blood Ketones >0.6 mmol/L - Algorithm 2
Description: as for outcome 13
Time Frame: 21 days
Measure: Number; unit: number of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 12 | 10
Number analyzed (Number of Mornings Analyzed) | 108 | 48
number of mornings | 3 | 1

15. Primary Outcome: Mornings With Blood Ketones >0.6 mmol/L - Algorithm 3
Description: as for outcome 13
Time Frame: 21 days
Measure: Number; unit: number of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 9 | 8
Number analyzed (Number of Mornings Analyzed) | 77 | 37
number of mornings | 1 | 0

16. Primary Outcome: Mornings With Urine Ketones Characterized as Moderate or Large - Algorithm 1
Description: The primary safety outcome will be evaluated by comparing the intervention and control nights and nights with vs. without actual shut-off of the pump for several measures of hyperglycemia such as number of mornings with urine ketones characterized as moderate or large based on measurement results of a urine dipstick test taken using Ketostix. Moderate is considered approximately 30 - 40 mg/dL and Large >80 mg/dL.
Time Frame: 21 days
Measure: Number; unit: number of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 5 | 5
Number analyzed (Number of Mornings Analyzed) | 67 | 38
number of mornings | 0 | 1

17. Primary Outcome: Mornings With Urine Ketones Characterized as Moderate or Large - Algorithm 2
Description: as for outcome 16
Time Frame: 21 days
Measure: Number; unit: number of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 12 | 10
Number analyzed (Number of Mornings Analyzed) | 108 | 48
number of mornings | 7 | 0

18. Primary Outcome: Mornings With Urine Ketones Characterized as Moderate or Large - Algorithm 3
Description: as for outcome 16
Time Frame: 21 days
Measure: Number; unit: number of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 9 | 8
Number analyzed (Number of Mornings Analyzed) | 77 | 37
number of mornings | 0 | 0

ADVERSE EVENTS:
Arm/Group | Predictive Pump Suspension Algorithm | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No